CLINICAL TRIAL: NCT03686878
Title: Safety and Efficacy of Lifitegrast 5% Ophthalmic Solution in Contact Lens Discomfort
Brief Title: Lifitegrast 5% Ophthalmic Solution and Contact Lens Dryness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EV Clinical Trials (Other)
Responsible Party: Principal Investigator, Agustin Gonzalez, Principal Investigator, EV Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LF5-CLD
Record Dates: First submitted 2018-09-18; First posted 2018-09-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Contact Lens; Contact Lens Discomfort; Contact Lens Dryness
Keywords: Keratoconjunctivitis Sicca; Dry Eye Disease; Eye Dryness
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes; Xerophthalmia | interventions — lifitegrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Group (Experimental): Lifitegrast 5% ophthalmic solution group
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Lifitegrast used twice a day

SUMMARY:
The most common reason for contact lens discontinuation is contact lens discomfort. The investigators believe that inflammation plays a role in contact lens discomfort and the use of lifitegrast 5% ophthalmic solution may reduce end of the day contact lens discomfort. This study will enroll 21 contact lens users who will be receiving lifitegrast 5% ophthalmic solution and monitor the contact lens discomfort for a 8 week period while.

DETAILED DESCRIPTION:
Contact lens discontinuation is mostly associated with ocular discomfort. Most patients identifying dryness as the primary reason for contact lens discontinuation. Patients often resort to contact lens solutions, lubricating and/or rewetting drops to temporality improve their contact lens wearing experience. Clinicians often resort to changing contact lens designs, solutions and wearing modalities to improve comfort.

Contact lens discomfort is believed to be mediated by many factors including inflammation and very similar in clinical symptoms of dry eye disease and symptoms of dryness.

Lifitegrast 5.0% ophthalmic solution is an FDA approved solution for the management of signs and symptoms of dryness of dry eye disease. Studies have shown lifitegrast 5% ophthalmic solution may work by blocking the interaction between ICAM-1 and LFA-1 leading to a decrease in activation and recruitment of T-cells, an initial step in inflammation.

The safety and efficacy of Xiidra has been studied in four, 12 week clinical trials involving over 2,100 patients for signs (https://www.xiidra-ecp.com/efficacy-treating-signs) and symptoms (https://www.xiidra-ecp.com/efficacy-symptom-improvement).

The purpose of this open label, interventional study is to examine the effect of lifitegrast 5% ophthalmic solution in contact lens wearing experience by using the CLDEQ-8.

ELIGIBILITY:
Inclusion Criteria:

1. Agree with study protocol
2. Provide Informed Consent
3. Age 21 or over
4. Previous 10 months history of self-assessed comfortable wear samfilcon A contact lenses

Exclusion Criteria:

1. Unable or unwilling to comply with study protocol
2. Unable of unwilling to provide Informed consent
3. Self-reported symptomatic intolerance of contact lenses
4. History of an active anterior segment, eyelids, eyelashes, corneal or conjunctival pathology, ongoing ocular infection, inflammation or any other ocular problem that would require management with additional topical ophthalmic medications.
5. Have had a history of corneal surgery (corneal transplants, LASIK, PRK).

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Change in CLDEQ-8 scores as reported by study participants | baseline to week 8
  measured changes in CLDEQ-8 scores as reported by study participants
Lisamine (corneal, conjunctiva) staining scores | baseline to week 8
  Lisamine score using the Oxford-Schema scoring

SECONDARY OUTCOMES:
Visual Acuity | Baseline to week 8
  Best corrected visual acuity measured by Snellen chart

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & Vision, Richardson, Texas, United States

REFERENCES:
- [Background] Efron N. Contact lens wear is intrinsically inflammatory. Clin Exp Optom. 2017 Jan;100(1):3-19. doi: 10.1111/cxo.12487. Epub 2016 Nov 2. PMID 27806431
- [Background] Godin MR, Gupta PK. Lifitegrast ophthalmic solution in the treatment of signs and symptoms of dry eye disease: design, development, and place in therapy. Clin Ophthalmol. 2017 May 22;11:951-957. doi: 10.2147/OPTH.S117188. eCollection 2017. PMID 28579745
- [Background] Nichols JJ, Willcox MD, Bron AJ, Belmonte C, Ciolino JB, Craig JP, Dogru M, Foulks GN, Jones L, Nelson JD, Nichols KK, Purslow C, Schaumberg DA, Stapleton F, Sullivan DA; members of the TFOS International Workshop on Contact Lens Discomfort. The TFOS International Workshop on Contact Lens Discomfort: executive summary. Invest Ophthalmol Vis Sci. 2013 Oct 18;54(11):TFOS7-TFOS13. doi: 10.1167/iovs.13-13212. No abstract available. PMID 24058135